CLINICAL TRIAL: NCT03605069
Title: A First in Human, Double-blind, Randomized, Intra-subject Placebo-controlled, Multiple Dose Study of QR-313 Evaluating Safety, Proof of Mechanism, Preliminary Efficacy and Systemic Exposure in Subjects With DDEB or RDEB Due to Mutation(s) in Exon 73 of the COL7A1 Gene
Brief Title: A Double-blind, Randomized, Intra-subject Placebo-controlled, Multicenter, Multiple Dose Study, Evaluating Safety, Proof of Mechanism, Preliminary Efficacy and Systemic Exposure in Subjects With Confirmed DDEB or RDEB Diagnosis With One or More Pathogenic Mutations in Exon 73 in the COL7A1 Gene
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Low enrollment
Sponsor: Phoenicis Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PQ-313-002; 2017-004806-17 (EudraCT Number)
Record Dates: First submitted 2018-06-25; First posted 2018-07-30 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Epidermolysis Bullosa Dystrophica, Recessive; Epidermolysis Bullosa Dystrophica, Dominant
Keywords: Recessive Dystrophic Epidermolysis Bullosa; EB; COL7A1; RNA Therapies; Antisense oligonucleotide; Exon skipping; WINGS; Topical treatment; RDEB; Exon 73; Mutations in exon 73; Dominant Dystrophic Epidermolysis Bullosa; DDEB
MeSH Terms: conditions — Epidermolysis Bullosa Dystrophica

STUDY DESIGN:
Intervention Model Description: intra-subject, placebo-controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- First TWA (A) (Other): In each subject up to two target wound areas (TWA) are randomized, one each to active treatment or placebo.
  In the first arm; randomization of the first selected TWA to active treatment or placebo
  Interventions: Drug: QR-313; Drug: Placebo
- Second TWA (B) (Other): In each subject, in the second arm; allocation of the second selected target wound area (TWA) to the alternative treatment. Second arm in the same subject as the first arm.
  Interventions: Drug: QR-313; Drug: Placebo

INTERVENTIONS:
Drug: QR-313 — QR-313 will be applied topically once daily for 8 weeks of treatment.
Drug: Placebo — Placebo will be applied topically once daily for 8 weeks of treatment.

SUMMARY:
A double-blind, randomized, intra-subject placebo-controlled, multicenter, multiple dose study, evaluating safety, proof of mechanism, preliminary efficacy and systemic exposure in subjects with confirmed DDEB or RDEB diagnosis with one or more pathogenic mutations in exon 73 in the COL7A1 gene.

DETAILED DESCRIPTION:
This clinical trial will evaluate the safety and tolerability, proof of mechanism, systemic exposure and preliminary efficacy following topical application of QR-313 to subjects with confirmed DDEB or RDEB with one or more pathogenic mutations in exon 73 in the COL7A1 gene.

Up to two Target Wound Areas (TWAs) per subject will be selected and randomized. Each TWA will be treated with IMP for 8 weeks, either QR-313 or matching placebo. All subjects will continue to be followed up for 8 weeks post last dose.

Subjects will be monitored through home visits and site visits. An imaging system will be used to assess the target wound at all home and study site visits.

QR-313 is a 21-nucleotide antisense oligonucleotide (AON) designed to hybridize to a specific sequence in the COL7A1 pre-messengerRNA (pre-mRNA).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, ≥ 4 years of age at Screening with a clinical diagnosis of DDEB or RDEB and at least one pathogenic mutation in exon 73 of the COL7A1 gene.
2. Have at least one TWA, ie, a skin area of 7 x 7 cm that ishows no signs of local infection, and contains a target wound that is either new or shows dynamic wound healing and complies to the following additional criteria:

   1. surface area of the target wound ranging from 5 to 30 cm2, located centrally in the selected 7 x 7 cm TWA.
   2. exposed sub-epidermal tissue to allow absorption of the IMP.
   3. no suspicion of current squamous cell carcinoma (SCC) upon visual inspection.

Exclusion Criteria:

1. Pregnant or breast-feeding female
2. Hemoglobin level at Screening requiring transfusion. The subject may be rescreened when the condition is considered stable.
3. Use of aminoglycosides, by any route of administration, except eye drops, 7 days or 5 half-lives, whichever is longer, prior to Baseline visit.
4. Untreated carcinoma of the TWA or history of carcinoma within 5 years prior to Screening, except adequately treated cutaneous squamous or basal cell carcinoma.
5. Life expectancy less than 6 months, as assessed by the Investigator
6. Current or known history of clinically significant hepatic or renal disease, that in the opinion of the Investigator, could impact subject safety or study participation.
7. Treatment with any systemic immunomodulators, immunosuppressants or cytotoxic chemotherapy within 2 months prior to the Baseline visit.
8. Use of any investigational drug or device within 28 days or 5 half-lives of the Baseline visit, whichever is longer, or plans to participate in another study of a drug or device during the study period. The washout of 5 half-lives does not apply to gene and cell therapy.
9. Known hypersensitivity to oligonucleotide treatment or excipients of the IMP.
10. Bleeding disorder or condition requiring the use of anticoagulants to be confirmed by aPTT by local lab within 48 hours of first treatment.
11. Use of systemic or topical steroids within 1 month prior to the baseline visit (inhaled and ophthalmic drops of corticosteroids or low dose topical solution of budesonide for esophagial strictures may be allowed).

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2018-07-02 (Actual); Primary Completion 2018-12-17 (Actual); Study Completion 2018-12-17 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment emergent adverse events/serious adverse events | through 8 weeks after last dose of IMP (EOS)
  Assessment of treatment emergent adverse events/serious adverse events
To assess the effect of QR-313 on the exclusion (skipping) of exon 73 from COL7A1 mRNA | after 4 weeks of treatment with IMP
  Absence of exon 73 in COL7A1 mRNA, detected by droplet digital polymerase chain reaction (ddPCR)

SECONDARY OUTCOMES:
Assessment of wound healing and skin strength measured in surface area (cm2) | through 8 weeks after last dose of IMP (EOS)
  Wound size (surface area in cm2)
Assessment of wound healing and skin strength as assessed by Physician Subjective Assessment of Severity (PSAS) | through 8 weeks after last dose of IMP (EOS)
  Wound severity as assessed by Physician Subjective Assessment of Severity (PSAS), a 3-point Likert static scale that classifies a wound in mild, moderate or severe
Assessment of wound healing and skin strength as assessed by Physician Subjective Assessment of Change (PSAC) | through 8 weeks after last dose of IMP (EOS)
  Wound change in severity as assessed by Physician Subjective Assessment of Change (PSAC), a 3-point Likert static scale that classifies a wound as mild, moderate or severe.
Assessment of wound healing and skin strength measuring onset of (re)blistering of a healed wound | through 8 weeks after last dose of IMP (EOS)
  Onset of (re)blistering of a healed wound
Assessment of wound healing and skin strength as assessed by Short Wound Specific Questionnaire (SWSQ) | through 8 weeks after last dose of IMP (EOS)
  Wound status as assessed by Short Wound Specific Questionnaire (SWSQ) addressing three domains: pruritus, pain, and inflammation. Pruritus and pain are recorded as a Patient Reported Outcome (PRO) measure. Inflammation is reported as an Observer Reported Outcome (ObsRO) measure.
Assessment of systemic exposure after topical administration of QR-313 to the target wound area (TWA) | Day 1 and after 4 and 8 weeks of treatment and EOS
  Serum levels of QR-313
Assessment of the effect of QR-313 on the presence of collagen type VII protein and anchoring fibrils | after 8 weeks of treatment
  Presence of collagen type VII protein expression (IIF microscopy)
Assessment of the effect of QR-313 on the presence of collagen type VII protein and anchoring fibrils | after 8 weeks of treatment
  Presence of anchoring fibrils (TEM)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Operations, Study Director — Phoenicis Therapeutics
Locations (6):
- United States (4):
  - Stanford University School of Medicine, LPCH, Palo Alto, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Journey Clinic, Center for Pediatric Blood and Marrow Transplantation, Minneapolis, Minnesota
  - Cincinnati Children's Hospital, Cincinnati, Ohio
- Hopital Necker Enfants Malades, Paris, France
- Hospital Universitario La Paz, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Miah KM, Hyde SC, Gill DR. Emerging gene therapies for cystic fibrosis. Expert Rev Respir Med. 2019 Aug;13(8):709-725. doi: 10.1080/17476348.2019.1634547. Epub 2019 Jun 27. PMID 31215818